CLINICAL TRIAL: NCT02049970
Title: Effect of the Addition of Dexmedetomidine to Bupivacaine During Supraclavicular Brachial Plexus Blockade for Forearm Surgery.
Brief Title: Effect of the Addition of Dexmedetomidine to Bupivacaine During Supraclavicular Brachial Plexus Blockade
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Recep Aksu, associate professor, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013/107
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Last update posted 2014-11-10 (Estimated); Status verified 2014-11

CONDITIONS: Sequelae of Fracture of Forearm and Upper Arm
Keywords: Supraclavicular block
MeSH Terms: interventions — Dexmedetomidine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- dexmedetomidine and bupivacaine (Experimental): Bupivacaine 50 mg and dexmedetomidine 1 microgram/kg
  Interventions: Drug: dexmedetomidine; Drug: bupivacaine
- Bupivacaine and placebo (Experimental): Bupivacaine 100 mg and SF 10 ml
  Interventions: Drug: dexmedetomidine; Drug: bupivacaine

INTERVENTIONS:
Drug: dexmedetomidine — 1 ml 100 mcg dexmedetomidine+ 15 ml 0.25 % bupivacaine are applied around brachial plexus
  Other Names: precedex
Drug: bupivacaine — 30 ml 0.25 % bupivacaine is applied around brachial plexus
  Other Names: marcaine

SUMMARY:
the aim of this study was effect of the addition of dexmedetomidine to bupivacaine during supraclavicular brachial plexus blockade for forearm surgery, by low doses bupivacaine providing prolonged analgesia after surgery.

DETAILED DESCRIPTION:
Anaesthesia for surgeries to the upper extremity commonly is provided using brachial plexus anaesthesia.Various local anaesthetic mixtures can be used to prolong local anaesthesia duration and epinephrine , opioids and dexmedetomidine are frequently used for this purpose. this study was conducted to compare the effects of adding dexmedetomidine to local anaesthetics in the supraclavicular brachial plexus block by using nerve stimulators and ultrasonography guided. dexmedetomidine has also been found the prolong the duration of bupivacaine infraclavicular brachial plexus block.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 age
* unwanted general anaesthesia
* ASA 1-2
* single forearm, arm surgery

Exclusion Criteria:

* major psychiatric problems
* major neurologic deficits
* coagulopathy
* drug allergies
* chronic analgesic used

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
the duration of sensorial block | postoperative 1 day
  pin-prick test

SECONDARY OUTCOMES:
the first time analgesic required | postoperative 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Recep Aksu, Study Director — Ass.Prof.
Locations (1):
- Erciyes University Medical Faculty, Kayseri, Turkey (Türkiye)